CLINICAL TRIAL: NCT04498728
Title: The Cardiac Acute Transitioning Care to Home (CATCH) Data Repository (CATCH App Repository)
Brief Title: Cardiac Acute Transitioning Care to Home (CATCH) App Data Repository
Acronym: CATCH
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Other Study IDs: Study00001436
Record Dates: First submitted 2020-07-30; First posted 2020-08-04 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Home Monitoring; Congenital Heart Disease; Mobile Health
Keywords: congenital heart disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Mobile Health Application for Remote Monitoring — The use of the CATCH application (CATCH App), and any data and images obtained from the use of the CATCH App, will all be performed as standard of care for patients at Children's Mercy Kansas City, and will be for the clinical treatment of patients. Data will be collected for the repository for all patients submitting data through the use of the CATCH App. Clinical care team will follow the patients after discharge home from the hospital.
  Other Names: CHAMP

SUMMARY:
This repository will consist of clinically derived data and images of patients with congenital heart disease from the time of birth until they have reached one of the following outcomes: transition to outpatient care that has not resulted in readmission in 30 days after hospital discharge, death, weaned off supplementary feeding tubes, or clinic visits demonstrating clinical stability with their primary cardiologist, or full bi-ventricular cardiac surgery palliation with improvement in hemodynamic stability. This information will be collected for clinical evaluation and diagnostic purposes and will continue to be stored for potential future research application.

DETAILED DESCRIPTION:
Approximately 40,000 infants are born each year with congenital heart disease (CHD), a leading cause of morbidity and mortality in infancy. Progress in surgical, transcatheter, and medical management of newborn CHD has significantly reduced mortality. The CHAMP app (separate IRB # 15030113) has helped to transition high-risk infants with single ventricle congenital heart disease out of the hospital and to second stage cardiac surgery at Children's Mercy Hospital and across the United States with improved survival. Remote monitoring technology and telemedicine is a critical tool to aid clinical care for high risk children with congenital heart disease but has been limited to the single ventricle population in most cases. The benefits of this tool as a standard of care for other children transitioning home may include decreased readmissions, improved weight gain, and remote monitoring for reduced throughput in the emergency room, hospital, and clinic settings. To improve outcomes beyond mortality and into morbidity with other high-risk patients with congenital heart disease, future studies must assess morbidities and quality of outcomes with the application of remote home monitoring with applications like the CHAMP app.

Patients that are discharging from the hospital after complex congenital heart disease surgery and cardiac catheterization are at high risk of events. Adverse outcomes in the year after discharge are of similar magnitude to mortality in hospital and are not only with infants with single ventricle heart disease but may include infants and children that were hospitalized more than 30 days, readmitted to intensive care unit more than once, smaller size for age, younger age at surgery, shunt dependent for pulmonary blood flow, congenital heart disease with complexities such as neurological conditions and supplemental enteral feedings gastrostomy. Over a 6-year period, 6.7% (514/7976) children experienced adverse events including mortality in a report from England after initial discharge from cardiac surgery. In a review of our similar patients from Children's Mercy we have noted a 5.8% mortality in this population.

There is additional focus on expanding transition care in the pediatric cardiac population beyond 30 days after discharge as traditionally followed by the Society of Thoracic Surgeons as a marker of well-state (traditionally 8.3%) and onto 90 days (21% of additional readmissions) to 1 year after discharge. Children had unplanned hospital readmissions during the first year after cardiac surgery that were between 31 and 90 days after discharge that could have possibly been prevented with the aid of remote technology in additional to ambulatory care by a specialized advanced practice nurse. Higher rates of readmissions were seen with those in lower socioeconomic areas (through zip codes), living closer to the hospital (potentially a marker of access to care and rurality), higher STAT category, longer intubation, and longer ICU length of stay were all markers for higher risk of later readmission after 31 days of discharge.

Combining the advancements with CHAMP app with the expert care teams with advanced practice nurses, a new standard of care for an expanded group of high-risk infants and children transitioning home after cardiac surgery and in-hospital care can be established. The research and ability to improve the understanding of how this process can be applied to an expanded population that has been identified as high risk is key for implementation and sustainability of a high risk transition care program.

ELIGIBILITY:
Inclusion Criteria:

* • Subjects with congenital heart disease that have been hospitalized for more than 30 days,

  * Subjects being discharged with readmissions more than twice to critical care areas,
  * Subject with single ventricle physiology that has not been discharged home during the single ventricle interstage period,
  * Subjects that are less than 18 years of age,
  * Subjects with gastrostomy or nasogastric tubes and congenital heart disease,
  * Subjects with congenital heart disease who are at a high risk for transition to the home setting and are not currently enrolled in the CHAMP single ventricle inclusion criteria, and/or
  * Subjects at high risk for events as identified by the Directors of the CATCH app Repository.

Exclusion Criteria:

* All patients not meeting at least one of the above specified criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children after hospitalization for heart surgery that required ICU care
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2021-05-29 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Number of children that had 30 day survival after hospital discharge | 1 month
  Survival of child after hospital discharge
Number of children that had Readmission after initiation hospital discharge | 2 months
  Hospital readmission after initial discharge

CONTACTS AND LOCATIONS:
Overall Officials: Lori Erickson, PhD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shirali G, Erickson L, Apperson J, Goggin K, Williams D, Reid K, Bradley-Ewing A, Tucker D, Bingler M, Spertus J, Rabbitt L, Stroup R. Harnessing Teams and Technology to Improve Outcomes in Infants With Single Ventricle. Circ Cardiovasc Qual Outcomes. 2016 May;9(3):303-11. doi: 10.1161/CIRCOUTCOMES.115.002452. Epub 2016 May 10. PMID 27166202
- [Result] Lushaj EB, Hermsen J, Leverson G, MacLellan-Tobert SG, Nelson K, Amond K, Anagnostopoulos PV. Beyond 30 Days: Analysis of Unplanned Readmissions During the First Year Following Congenital Heart Surgery. World J Pediatr Congenit Heart Surg. 2020 Mar;11(2):177-182. doi: 10.1177/2150135119895212. PMID 32093562
- [Result] Bingler M, Erickson LA, Reid KJ, Lee B, O'Brien J, Apperson J, Goggin K, Shirali G. Interstage Outcomes in Infants With Single Ventricle Heart Disease Comparing Home Monitoring Technology to Three-Ring Binder Documentation: A Randomized Crossover Study. World J Pediatr Congenit Heart Surg. 2018 May;9(3):305-314. doi: 10.1177/2150135118762401. PMID 29692236